CLINICAL TRIAL: NCT05989672
Title: A Phase 1, Observer-blind, Randomized, Placebo-Controlled Study to Evaluate Reactogenicity, Safety and Immune Response of an HSV-targeted Immunotherapy in HSV-2 Seronegative Japanese Participants Aged 18-40 Years
Brief Title: A Study on the Reactogenicity, Safety and Immune Response of a Targeted Immunotherapy Against HSV in Healthy Japanese Participants Aged 18-40 Years
Acronym: TH HSV REC-004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 218459
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Herpes Simplex
Keywords: Herpes Simplex Virus genital herpes; Herpes Simplex Virus; Reactogenicity; Safety; Immune response
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Herpes Simplex Virus (HSV)-Targeted Immunotherapy (HSVTI)_Formulation 1 (F1) group (Experimental): HSV-2 seronegative participants received HSVTI Formulation 1 (high dose) as the study intervention at Day 1 and Day 29.
  Interventions: Biological: HSVTI Formulation 1
- HSVTI_Formulation 2 (F2) group (Experimental): HSV-2 seronegative participants received HSVTI Formulation 2 (low dose) as the study intervention at Day 1 and Day 29.
  Interventions: Biological: HSVTI Formulation 2
- Placebo group (Placebo Comparator): HSV-2 seronegative participants received placebo as control at Day 1 and Day 29.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HSVTI Formulation 1 — This investigational intervention was administered intramuscularly to HSVTI_F1 Group.
  Arms: Herpes Simplex Virus (HSV)-Targeted Immunotherapy (HSVTI)_Formulation 1 (F1) group
Biological: HSVTI Formulation 2 — This investigational intervention was administered intramuscularly to HSVTI_F2 Group.
  Arms: HSVTI_Formulation 2 (F2) group
Biological: Placebo — This intervention was administered intramuscularly to Placebo group.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of 2 formulations of Herpes Simplex Virus (HSV)-Targeted Immunotherapy (HSVTI) in HSV-2 seronegative ethnic Japanese adults aged 18-40 years.

ELIGIBILITY:
Inclusion Criteria:

• Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).

* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants as established by medical history and physical examination, at the discretion of the investigator, before entering into the study.
* Man or woman aged 18 to 40 years, included, at the time of screening.
* Japanese ethnic origin (defined as having been born in Japan with 4 ethnic Japanese grandparents and able to speak Japanese).
* Women of non-childbearing potential may be enrolled in the study.
* Women of childbearing potential may be enrolled in the study, if the participant:

  * Has practiced highly effective contraception for 1 month prior to study intervention administration, and
  * Has a negative pregnancy test result at the Screening visit and on the day of each study intervention administration, and
  * Has agreed to continue highly effective contraception until Day 118, approximately 3 months post-Dose 2.

Blood sample for simultaneous FSH and estradiol levels may be collected and tested locally at the discretion of the investigator to confirm non-reproductive potential according to local laboratory reference range.

• Seronegative for HSV-2 as determined by Western blot performed at the Screening visit.

Exclusion Criteria:

Medical conditions:

* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, endocrine, or renal functional abnormality, as determined by physical examination or laboratory screening tests.

  * Clinically significant abnormalities may include but are not limited to: evidence of cardiac damage, heart failure categorized as class II or greater according to the New York Heart Association functional classification, heart valve disease, pulmonary uncontrolled persistent asthma despite treatment, uncontrolled diabetes, or disease or disorder that may put the participant at risk or influence study results.
  * Participants with a controlled underlying chronic co-morbidity may be enrolled, provided there have been no changes to their medication within 3 months prior to the Screening visit.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study or that would interfere with the immunogenicity assessments planned in this study.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Any confirmed or suspected immunosuppressive or immunodeficient condition or documented or suspected HIV infection, based on medical history and physical examination (no laboratory testing required).

Hypersensitivity to latex.

* Recurrent history of or uncontrolled neurological disorders or seizures.
* At the screening visit: hematological parameters (hemoglobin level, white blood cell, platelet) and/or biochemical parameters (ALT, AST, creatinine, blood urea nitrogen) outside the normal laboratory ranges, unless the laboratory abnormalities are considered not clinically significant by the investigator.
* Body mass index =18 kg/m2 or =35 kg/m2.
* History of any form of ocular HSV infection, HSV-related erythema multiforme, or HSV-related neurological complications (including meningitis, encephalitis, radiculopathy, myelitis).

Prior/Concomitant therapy:

* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study intervention during the period beginning as of the Screening visit, or their planned use during the study period.
* Planned administration or administration of a vaccine* in the period starting 15 days* before each dose and ending 15 days* after each dose of study intervention administration**.

  * In case of adjuvanted and live-attenuated vaccines, this time window is to be increased to 30 days before and after each dose.
  * In case emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced if, necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.
* Administration or planned administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first dose of study intervention or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose. For corticosteroids, this will mean prednisone equivalent =20 mg/day for adult participants. Inhaled, intra articular and topical steroids are allowed.
* Prior receipt of a vaccine containing HSV antigens.

Prior/Concurrent clinical study experience:

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug or invasive medical device).

Other exclusions:

• Pregnant or lactating woman. Woman planning to become pregnant or planning to discontinue contraceptive precautions before Day 118 (approximately 3 months post-Dose 2).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Groups:
- Herpes Simplex Virus (HSV)-Targeted Immunotherapy (HSVTI)_F1 Group: HSV-2 seronegative participants received HSVTI Formulation 1 (high dose) as the study intervention at Day 1 and Day 29.
- HSVTI_F2 Group: HSV-2 seronegative participants received HSVTI Formulation 2 (low dose) as the study intervention at Day 1 and Day 29.
Period: Overall Study
Arm/Group | Herpes Simplex Virus (HSV)-Targeted Immunotherapy (HSVTI)_F1 Group | HSVTI_F2 Group | Placebo Group
Started | 20 | 20 | 10
Completed | 17 | 20 | 10
Not Completed | 3 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HSVTI_F1 Group: HSV-2 seronegative participants received HSVTI Formulation 1 (high dose) as the study intervention at Day 1 and Day 29.
- Total: Total of all reporting groups
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group | Total
Number analyzed (Participants) | 20 | 20 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 29.9 (8.0) | 27.2 (6.7) | 31.4 (6.6) | 29.1 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 6 | 28
  Male | 9 | 9 | 4 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - JAPANESE HERITAGE | 20 | 20 | 10 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Events
Description: The solicited administration site events include erythema (redness), pain and swelling. Any solicited administration site AEs = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 1
Population: Analysis was performed on the Exposed set (ES), which included all participants who received at least one dose of the study intervention and have post-vaccination data for the specified analysis at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Erythema | 8 | 2 | 0
  Pain | 19 | 18 | 4
  Swelling | 4 | 3 | 0

2. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Events
Description: as for outcome 1
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 29
Population: Analysis was performed on the ES. Only participants with data available at specified timepoints were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 17 | 20 | 10
Participants
  Erythema | 2 | 4 | 0
  Pain | 15 | 14 | 0
  Swelling | 4 | 2 | 0

3. Primary Outcome: Number of Participants Reporting Any Solicited Systemic Events
Description: The solicited systemic events include arthralgia (joint pain), fatigue (tiredness), headache, myalgia (muscle pain), and fever [temperature >=38.0-degree Celsius (°C)]. Any solicited systemic AEs = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Arthralgia | 6 | 5 | 0
  Fatigue | 16 | 6 | 1
  Headache | 10 | 5 | 2
  Myalgia | 11 | 8 | 1
  Fever | 3 | 1 | 0

4. Primary Outcome: Number of Participants Reporting Any Solicited Systemic Events
Description: The solicited systemic events include arthralgia (joint pain), fatigue (tiredness), headache, myalgia (muscle pain), and fever (temperature >= 38.0 °C). Any solicited systemic AEs = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7 days (including the day of vaccination) following vaccination at Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 17 | 20 | 10
Participants
  Arthralgia | 6 | 4 | 0
  Fatigue | 13 | 7 | 1
  Headache | 7 | 2 | 1
  Myalgia | 9 | 5 | 0
  Fever | 5 | 0 | 0

5. Primary Outcome: Number of Participants Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is an AE that was not included in the list of solicited events. Also, any solicited symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited AE. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 28 days (including the day of vaccination) following vaccination at Day 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 4 | 4 | 4

6. Primary Outcome: Number of Participants Reporting Any Unsolicited AEs
Description: as for outcome 5
Time Frame: During the 28 days (including the day of vaccination) following vaccination at Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 17 | 20 | 10
Participants | 4 | 3 | 2

7. Primary Outcome: Number of Participants Reporting Any Medically Attended Events (MAEs)
Description: MAEs are defined as AEs requiring medically attended visits, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: From Day 1 (dose 1) up to Day 57 (28 days post dose 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 1 | 1 | 3

8. Primary Outcome: Number of Participants Reporting Any Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: From Day 1 (dose 1) up to Day 57 (28 days post dose 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 0 | 0 | 0

9. Primary Outcome: Number of Participants Reporting Any Newly Diagnosed Potential Immune-Mediated Diseases (pIMDs)
Description: plMDs are defined as a subset of adverse events of special interest (AESI) that include autoimmune diseases and other inflammatory or neurologic disorders that may or may not have an autoimmune etiology. Newly diagnosed pIMDs are categorized as new-onset conditions if they start following the administration of the study intervention. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: From Day 1 (dose 1) up to Day 57 (28 days post dose 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 0 | 0 | 0

10. Primary Outcome: Number of Participants Reporting Any Exacerbation of Pre-existing pIMDs
Description: Exacerbation of pre-existing pIMDs is categorized as an exacerbation of a pre-existing chronic condition if the condition worsened following the administration of the study intervention.
Time Frame: From Day 1 (dose 1) up to Day 57 (28 days post dose 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 0 | 0 | 0

11. Primary Outcome: Number of Participants Reporting Any Hematological and Biochemical Laboratory Abnormalities
Description: The safety laboratory data included haematological parameters (hemoglobin, white blood cells (WBC), platelets), and chemical parameters (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], Creatinine, Urea nitrogen). Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 1 (pre-study intervention administration)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants
  ALT: Below | 0 | 0 | 0
  ALT: Within | 20 | 20 | 10
  ALT: Above | 0 | 0 | 0
  AST: Below | 0 | 0 | 0
  AST: Within | 20 | 20 | 10
  AST: Above | 0 | 0 | 0
  Creatinine: Below | 0 | 0 | 0
  Creatinine: Within | 20 | 20 | 10
  Creatinine: Above | 0 | 0 | 0
  Urea Nitrogen: Below | 2 | 2 | 2
  Urea Nitrogen: Within | 18 | 18 | 8
  Urea Nitrogen: Above | 0 | 0 | 0
  Hemoglobin: Below | 8 | 3 | 2
  Hemoglobin: Within | 12 | 17 | 8
  Hemoglobin: Above | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0
  Platelets: Within | 20 | 20 | 10
  Platelets: Above | 0 | 0 | 0
  WBC: Below | 0 | 1 | 0
  WBC: Within | 19 | 19 | 10
  WBC: Above | 1 | 0 | 0

12. Primary Outcome: Number of Participants Reporting Any Hematological and Biochemical Laboratory Abnormalities
Description: as for outcome 11
Time Frame: At Day 8 (7 days post dose 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants
  ALT: Below | 0 | 0 | 0
  ALT: Within | 20 | 19 | 10
  ALT: Above | 0 | 1 | 0
  AST: Below | 0 | 0 | 0
  AST: Within | 20 | 20 | 10
  AST: Above | 0 | 0 | 0
  Creatinine: Below | 1 | 0 | 0
  Creatinine: Within | 19 | 20 | 10
  Creatinine: Above | 0 | 0 | 0
  Urea Nitrogen: Below | 2 | 1 | 2
  Urea Nitrogen: Within | 18 | 18 | 8
  Urea Nitrogen: Above | 0 | 1 | 0
  Hemoglobin: Below | 6 | 5 | 2
  Hemoglobin: Within | 14 | 15 | 8
  Hemoglobin: Above | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0
  Platelets: Within | 20 | 20 | 10
  Platelets: Above | 0 | 0 | 0
  WBC: Below | 0 | 2 | 1
  WBC: Within | 20 | 18 | 9
  WBC: Above | 0 | 0 | 0

13. Primary Outcome: Number of Participants Reporting Any Hematological and Biochemical Laboratory Abnormalities
Description: as for outcome 11
Time Frame: At Day 29 (28 days post dose 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 17 | 20 | 10
Participants
  ALT: Below | 0 | 0 | 0
  ALT: Within | 17 | 19 | 10
  ALT: Above | 0 | 1 | 0
  AST: Below | 0 | 0 | 0
  AST: Within | 17 | 20 | 10
  AST: Above | 0 | 0 | 0
  Creatinine: Below | 1 | 0 | 0
  Creatinine: Within | 16 | 20 | 10
  Creatinine: Above | 0 | 0 | 0
  Urea Nitrogen: Below | 1 | 1 | 1
  Urea Nitrogen: Within | 16 | 19 | 9
  Urea Nitrogen: Above | 0 | 0 | 0
  Hemoglobin: Below | 9 | 5 | 2
  Hemoglobin: Within | 8 | 15 | 8
  Hemoglobin: Above | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0
  Platelets: Within | 17 | 20 | 10
  Platelets: Above | 0 | 0 | 0
  WBC: Below | 1 | 1 | 0
  WBC: Within | 15 | 19 | 10
  WBC: Above | 1 | 0 | 0

14. Primary Outcome: Number of Participants Reporting Any Hematological and Biochemical Laboratory Abnormalities
Description: as for outcome 11
Time Frame: At Day 36 (7 days post dose 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 17 | 20 | 10
Participants
  ALT: Below | 0 | 0 | 0
  ALT: Within | 17 | 19 | 10
  ALT: Above | 0 | 1 | 0
  AST: Below | 0 | 0 | 0
  AST: Within | 17 | 20 | 10
  AST: Above | 0 | 0 | 0
  Creatinine: Below | 2 | 0 | 1
  Creatinine: Within | 15 | 20 | 9
  Creatinine: Above | 0 | 0 | 0
  Urea Nitrogen: Below | 1 | 2 | 0
  Urea Nitrogen: Within | 15 | 18 | 10
  Urea Nitrogen: Above | 1 | 0 | 0
  Hemoglobin: Below | 6 | 4 | 2
  Hemoglobin: Within | 11 | 16 | 8
  Hemoglobin: Above | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0
  Platelets: Within | 17 | 20 | 10
  Platelets: Above | 0 | 0 | 0
  WBC: Below | 2 | 2 | 0
  WBC: Within | 14 | 18 | 10
  WBC: Above | 1 | 0 | 0

15. Primary Outcome: Number of Participants Reporting Any Hematological and Biochemical Laboratory Abnormalities
Description: as for outcome 11
Time Frame: At Day 57 (28 days post dose 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 17 | 20 | 10
Participants
  ALT: Below | 0 | 0 | 0
  ALT: Within | 17 | 20 | 10
  ALT: Above | 0 | 0 | 0
  AST: Below | 0 | 0 | 0
  AST: Within | 17 | 20 | 10
  AST: Above | 0 | 0 | 0
  Creatinine: Below | 2 | 2 | 0
  Creatinine: Within | 15 | 18 | 10
  Creatinine: Above | 0 | 0 | 0
  Urea Nitrogen: Below | 3 | 1 | 1
  Urea Nitrogen: Within | 14 | 18 | 8
  Urea Nitrogen: Above | 0 | 1 | 1
  Hemoglobin: Below | 8 | 6 | 1
  Hemoglobin: Within | 9 | 14 | 9
  Hemoglobin: Above | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0
  Platelets: Within | 17 | 20 | 10
  Platelets: Above | 0 | 0 | 0
  WBC: Below | 1 | 2 | 0
  WBC: Within | 16 | 18 | 10
  WBC: Above | 0 | 0 | 0

16. Secondary Outcome: Percentage of Participants With Seropositivity Rate of Anti-HSVTI Antibody
Description: The seropositivity rate of anti-HSVTI antibody was assessed by Enzyme-Linked Immunosorbent Assay (ELISA) and measured in ELISA Units per milliliter (EU/mL).
Time Frame: At Day 1 (pre-study intervention administration), Day 29 (28 days post-Dose 1), and Day 57 (28 days post-Dose 2)
Population: Analysis was performed on the Per Protocol set for analysis of humoral immunogenicity (PPS_Immuno) which included all participants who received all doses as per protocol, have immunogenicity results post-dose, complied with dosing/blood draw intervals, without intercurrent conditions that may interfere with immunogenicity, without prohibited concomitant medication/vaccination and have post-vaccination data for the specified analysis at specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Percentage of participants
  Day 1 | 20.0 [5.7 to 43.7] | 25.0 [8.7 to 49.1] | 20.0 [2.5 to 55.6]
  Day 29: number analyzed (Participants) | 17 | 20 | 10
  Day 29 | 100 [80.5 to 100.0] | 100 [83.2 to 100.0] | 20.0 [2.5 to 55.6]
  Day 57: number analyzed (Participants) | 17 | 20 | 10
  Day 57 | 100 [80.5 to 100.0] | 100 [83.2 to 100.0] | 20.0 [2.5 to 55.6]

17. Secondary Outcome: Anti-HSVTI Antibody Geometric Mean Concentration (GMC)
Time Frame: At Day 1 (pre-study intervention administration), Day 29 (28 days post-Dose 1), and Day 57 (28 days post-Dose 2)
Population: Analysis was performed on the PPS_Immuno. Only participants with data available at specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
EU/mL
  Day 1 | 1.2 [0.5 to 2.8] | 1.0 [0.5 to 2.0] | 1.1 [0.3 to 3.5]
  Day 29: number analyzed (Participants) | 17 | 20 | 10
  Day 29 | 270.1 [176.5 to 413.4] | 197.8 [134.6 to 290.7] | 1.1 [0.3 to 3.8]
  Day 57: number analyzed (Participants) | 17 | 20 | 10
  Day 57 | 558.8 [331.4 to 942.2] | 390.8 [221.9 to 688.3] | 1.1 [0.3 to 4.0]

18. Secondary Outcome: Geometric Mean of HSVTI-specific Cluster of Differentiation (CD)4+T Cells Frequency
Description: The geometric mean of HSVTI CD4+T cells frequency expressing at least 2 markers including at least one cytokine among Interferon [IFN]-gamma, Tumour necrosis factor [TNF]-alpha, Interleukin [IL]-2, IL-13, IL-17, 4-1BB and CD40L were assessed by Intracellular staining (ICS).
Time Frame: At Day 1 (pre-study intervention administration), Day 29 (28 days post-Dose 1), and Day 57 (28 days post-Dose 2)
Population: Analysis was performed on the Per Protocol set for analysis of cellular immunogenicity (PPS_CMI) which included all participants who received all doses as per protocol, have CMI results post-dose, complied with dosing/blood draw intervals, without intercurrent conditions that may interfere with immunogenicity, without prohibited concomitant medication/vaccination and have post-vaccination data for the specified analysis at specified timepoints.
Measure: Geometric Mean (Standard Deviation); unit: HSVTI-specifc CD4+ T cells/10^6 cells
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 19 | 20 | 10
HSVTI-specifc CD4+ T cells/10^6 cells
  Day 1: number analyzed (Participants) | 19 | 18 | 10
  Day 1 | 64.0 (0.9) | 36.3 (1.0) | 24.0 (0.9)
  Day 29: number analyzed (Participants) | 15 | 20 | 10
  Day 29 | 456.8 (0.5) | 199.1 (0.8) | 21.1 (1.1)
  Day 57: number analyzed (Participants) | 16 | 19 | 10
  Day 57 | 5899.7 (0.4) | 2932.3 (0.4) | 40.3 (1.0)

19. Secondary Outcome: Geometric Mean of HSVTI-specific CD8+ T Cells Frequency
Description: The geometric mean of HSVTI CD8+ T cells frequency expressing at least 2 activation markers including at least one cytokine among IFN-gamma, TNF-alpha, IL-2, IL-13, IL- 17, 4-1BB and CD40L were assessed by ICS.
Time Frame: At Day 1 (pre-study intervention administration), Day 29 (28 days post-Dose 1), and Day 57 (28 days post-Dose 2)
Population: Analysis was performed on the PPS_CMI. Only participants with data available at specified timepoints were included in the analysis.
Measure: Geometric Mean (Standard Deviation); unit: HSVTI-specifc CD8+ T cells/10^6 cells
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 19 | 20 | 10
HSVTI-specifc CD8+ T cells/10^6 cells
  Day 1: number analyzed (Participants) | 19 | 18 | 10
  Day 1 | 37.6 (0.8) | 19.6 (0.9) | 8.7 (0.8)
  Day 29: number analyzed (Participants) | 16 | 20 | 10
  Day 29 | 27.1 (1.0) | 9.5 (0.8) | 8.6 (0.7)
  Day 57: number analyzed (Participants) | 17 | 19 | 10
  Day 57 | 61.0 (0.9) | 20.8 (0.8) | 13.5 (0.9)

20. Secondary Outcome: Number of Participants Reporting Any MAEs
Time Frame: From Day 1 (dose 1) up to study end (Day 209)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 3 | 1 | 4

21. Secondary Outcome: Number of Participants Reporting Any SAEs
Time Frame: From Day 1 (dose 1) up to study end (Day 209)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 0 | 0 | 0

22. Secondary Outcome: Number of Participants Reporting Any Newly Diagnosed pIMDs
Time Frame: From Day 1 (dose 1) up to study end (Day 209)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 0 | 0 | 0

23. Secondary Outcome: Number of Participants Reporting Any Exacerbation of Pre-existing pIMDs
Time Frame: From Day 1 (dose 1) up to study end (Day 209)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 10
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs: during the 7-day follow-up period after any vaccination. Unsolicited AEs: during the 28-day follow-up period after any vaccination. All- cause mortality, SAEs, MAEs and plMDs (newly diagnosed and pre-existing pIMDs): from first vaccination (Day 1) up to study end (Day 209)
Arm/Group | HSVTI_F1 Group | HSVTI_F2 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSVTI_F1 Group (N=20) | HSVTI_F2 Group (N=20) | Placebo Group (N=10)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental abfraction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary gland pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Administration site erythema (General disorders) | 9 (10) | 4 (6) | 0 (0)
Administration site pain (General disorders) | 19 (35) | 19 (32) | 4 (4)
Administration site pruritus (General disorders) | 1 (1) | 2 (3) | 0 (0)
Administration site swelling (General disorders) | 5 (8) | 4 (6) | 0 (0)
Chills (General disorders) | 3 (3) | 2 (2) | 0 (0)
Fatigue (General disorders) | 18 (29) | 10 (13) | 1 (2)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (12) | 5 (9) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (20) | 8 (13) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 12 (17) | 6 (7) | 2 (3)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT05989672/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT05989672/SAP_001.pdf